CLINICAL TRIAL: NCT03127722
Title: An Open-label, Non-randomized, Prospective Observational Cohort Study to Assess Post-procedural Outcomes in Two Cohorts of Women Who Chose to Undergo Either Hysteroscopic Sterilization (Essure®) or Laparoscopic Tubal Sterilization
Brief Title: Study to Assess Outcomes in Women Undergoing Either Hysteroscopic Sterilization (Essure®) or Laparoscopic Tubal Sterilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18894
Record Dates: First submitted 2017-03-05; First posted 2017-04-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Contraception
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ESSURE (BAY1454032) (Experimental): Subjects selecting hysteroscopic sterilization who are not contraindicated for the Essure procedure according to the most current approved version of the Essure IFU. Subject willing to use alternative contraception for at least 3 months post-Essure placement procedure, until a satisfactory Essure Confirmation Test is documented.
  Interventions: Procedure: Blood draw; Device: ESSURE (BAY1454032)
- Laparoscopic tubal sterilization (Active Comparator): Subjects selecting laparoscopic sterilization who are not contraindicated for laparoscopic tubal sterilization according to common clinical practice standard of care
  Interventions: Procedure: Blood draw; Procedure: Laparoscopic tubal sterilization

INTERVENTIONS:
Procedure: Blood draw — Decision for either treatment will be based upon clinical practice and physician/patient counseling. In addition of routine care practice, blood draws will be performed at baseline, 12 months and 60 months on subjects undergoing either an ESSURE procedure or a laparoscopic tubal sterilization.
Device: ESSURE (BAY1454032) — Decision for either treatment will be based upon clinical practice and physician/patient counseling, and will not be specified in the study protocol.
  Arms: ESSURE (BAY1454032)
Procedure: Laparoscopic tubal sterilization — Decision for either treatment will be based upon clinical practice and physician/patient counseling, and will not be specified in the study protocol.
  Arms: Laparoscopic tubal sterilization

SUMMARY:
This study is designed to assess post-procedural outcomes for women who chose to undergo either hysteroscopic sterilization (Essure®) or laparoscopic tubal sterilization, including:

* Pelvic and/or lower abdominal pain
* Abnormal uterine bleeding
* Surgical intervention (including "insert removal" and hysterectomy)
* Allergic, hypersensitivity, or autoimmune-like reactions

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 21 years of age;
* Subjects of all weights will be included;
* Subjects who are scheduled to undergo an Essure insert placement procedure for permanent birth control or laparoscopic tubal sterilization. Decision for either treatment based upon clinical practice and physician/patient counseling.
* For the Essure group only:

  • Subjects selecting hysteroscopic sterilization who are not contraindicated for the Essure procedure according to the most current approved version of the Essure IFU;
* For the laparoscopic tubal sterilization group only:

  * Subjects selecting laparoscopic sterilization who are not contraindicated for laparoscopic tubal sterilization according to common clinical practice standard of care.

Exclusion Criteria:

* Subjects who are post-menopausal;
* Subjects suspected of being or confirmed pregnant;
* Subjects post-partum or undergone pregnancy termination ≤6 weeks prior to scheduled procedure;
* Subjects uncertain about ending fertility;
* Subjects with an active upper or lower genital tract infection;
* Subjects with gynecologic malignancy (suspected or known);
* Subjects who have had an attempted prior sterilization procedure (either laparoscopic or hysteroscopic);
* Subjects scheduled to undergo concomitant intrauterine or laparoscopic procedures at the time of insert placement (intrauterine device removal is not considered a concomitant procedure) or laparoscopic sterilization;
* Subjects with unexplained vaginal bleeding.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain: The proportion of AEs of chronic lower abdominal and/or pelvic pain after insertion of Essure System compared to the proportion of AEs of chronic lower abdominal and/or pelvic pain after laparoscopic tubal sterilization | Up to 60 months
  All AEs will be assessed and documented by the investigator according to seriousness, intensity, action taken, treatments, outcome and causal relationship.
Bleeding: The proportion of AEs of abnormal uterine bleeding (AUB) after insertion of Essure System compared to the proportion of AEs of AUB after laparoscopic tubal sterilization | Up to 60 months
  All AEs will be assessed and documented by the investigator according to seriousness, intensity, action taken, treatments, outcome and causal relationship.
Hypersensitivity / allergy / autoimmune disorders: The proportion of subjects with new onset or worsening allergic/hypersensitivity reactions and newly diagnosed or worsening autoimmune disorders in Essure vs laparoscopic tubal sterilization arms | Up to 60 months
  All AEs will be assessed and documented by the investigator according to seriousness, intensity, action taken, treatments, outcome and causal relationship.
Proportion of subjects undergoing invasive gynecologic surgery after Essure placement (excluding second placement attempts), including Essure removal compared to subjects undergoing invasive gynecologic surgery after laparoscopic tubal sterilization | Up to 60 months
  All AEs will be assessed and documented by the investigator according to seriousness, intensity, action taken, treatments, outcome and causal relationship.
Patient reported outcomes for health status | Up to 60 months
  Medical Outcomes Study Short Form-36
Patient reported outcomes for pain intensity | Up to 60 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) scale V1.0, form ´Pain Intensity 3a´. Pain intensity is assessed via questions and ranked across 5 levels from ´No pain´ to ´Very severe pain´.
Patient reported outcomes for pain interference | Up to 60 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) scale V1.0, form ´Pain Interference 8a´. Pain interference is assessed via questions and ranked across 5 levels from ´Not at all´ to ´Very much´.
Patient reported outcomes for bleeding by AMSS | Up to 60 months
  Aberdeen Menorrhagia Severity Scale (AMSS) is used to characterize bleeding. AMSS is a questionaire consisting of 13 items giving a total score from 0 (least severe) to 42 points (most severe).
Patient reported outcomes for bleeding by intermenstrual bleeding questions | Up to 60 months
  Two questions used to characterize intermenstrual bleeding.
Patient reported outcomes for centralized pain | At baseline
  Assessed with the Fibromyalgia Survey Questionnaire
Patient reported outcomes on adverse events from device reports | Up to 60 months
  Assessed by questionnaires to actively solicit information on adverse events found in medical device reporting (MDR) reports with Essure and control potential bias in adverse event reporting.
Patient reported outcomes on media sources for their medical decisioning | Up to 60 months
  Assessed by Social Media questionnaire to elicit information about sources of influence on medical decisions.
Rates of AEs in subjects undergoing Essure placement and laparoscopic tubal sterilization | Up to 60 months
  All AEs will be assessed and documented by the investigator according to seriousness, intensity, action taken, treatments, outcome and causal relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (57):
- United States (57):
  - New Horizons Women's Care, Chandler, Arizona
  - Precision Trials, AZ, LLC, Phoenix, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - United Clinical Research, Huntington Beach, California
  - Orange Coast Women's Medical Group - Laguna Hills Office, Laguna Hills, California
  - Physicians Research Options, LLC, Lakewood, Colorado
  - The Women's Health Group, P.C., Thornton, Colorado
  - M & O Clinical Research, LLC, Fort Lauderdale, Florida
  - Altus Research, Lake Worth, Florida
  - Universal Axon Clinical Research, Miami, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Clinical Research Prime, LLLP, Idaho Falls, Idaho
  - John H Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Women's Health Advantage, Fort Wayne, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - Office of Dr. Cindy Basinski, LLC, Newburgh, Indiana
  - Women's Health Care, PC, Newburgh, Indiana
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - University of Kentucky Albert B. Chandler Hospital, Lexington, Kentucky
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - Mid-Atlantic Permanente Research Institute, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Women's Integrated Health Care, PC, Grand Blanc, Michigan
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Columbia University Medical Center, New York, New York
  - Unified Women's Clinical Research, LLC, Greensboro, North Carolina
  - Women's Health Alliance, Raleigh, North Carolina
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Seven Hills Women's Health Centers, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Columbus OB-GYN/Radiant Research, Columbus, Ohio
  - Complete Healthcare for Women, Inc., Columbus, Ohio
  - Wright State Physicians Health Center, Dayton, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - HillTop Obstetrics & Gynecology, Franklin, Ohio
  - Amy Brenner, MD & Associates, LLC, Mason, Ohio
  - AC Clinical Research, Tiffin, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's Hospital - Allentown Campus, Allentown, Pennsylvania
  - Women's Health Care Group of PA, Pottstown, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women & Infants Hospital (OGCC), Providence, Rhode Island
  - Palmetto Clinical Research (PCR), Charleston, South Carolina
  - OB-GYN Centre of Excellence, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Ben Taub General Hospital, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - Southeast Texas Family Planning and Cancer Screening, Houston, Texas
  - Brown Stone Clinical Trials, LLC, Irving, Texas
  - Tanner Clinic, Layton, Utah
  - Women's Healthcare Associates, LLC - Tualatin, Pleasant Grove, Utah
  - Tidewater Clinical Research, Inc., Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/18894